CLINICAL TRIAL: NCT04968821
Title: Telehealth Physical Activity Intervention After Lumbar Spine Surgery
Brief Title: Telehealth Activity Intervention After Lumbar Spine Surgery
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Academy of Orthopaedic Physical Therapy (Unknown)
Responsible Party: Principal Investigator, Kristin Archer, Professor, Department of Orthopaedics & Rehab, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211126
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Spinal Degenerative Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Participants randomized to the physical activity intervention will receive usual postoperative care and a tele-health physical activity intervention.
  Interventions: Behavioral: Physical activity intervention
- Usual Care (Other): Participants randomized to usual care will receive postoperative care as determined by their treating surgeon.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Physical activity intervention — Participants randomized to the physical activity intervention will receive a Fitbit and be enrolled in Fitabase (Fitbit tracking system). Participants will also participate in 8 tele-health sessions with a physical therapist. Sessions will involve setting weekly physical activity goals and reviewing the participant's physical activity on the Fitbit tracking system.
  Arms: Physical Activity
Other: Usual care — Usual postoperative care includes surgeon-directed lifting restrictions, advice to stay active, and oral analgesics as needed. Physical therapy referral will be at the discretion of the surgeon. However, physical therapy is not typically started until 12 weeks after surgery.
  Arms: Usual Care

SUMMARY:
The overall objective of this randomized controlled study is to examine the preliminary efficacy of a physical activity intervention that includes wearable technology and remote physical therapist support in patients undergoing lumbar spine surgery. Patients will be randomized to receive 8 sessions of a telehealth physical activity intervention (n=30) or usual postoperative care (n=30). The Investigator's central hypothesis is that a postoperative telehealth physical activity intervention will lead to greater improvements in objective physical activity (primary outcome) and patient-reported physical function, disability, and pain (secondary outcomes) compared to usual care in patients undergoing lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years or older
2. Scheduled for surgical treatment of a lumbar degenerative condition using laminectomy with or without arthrodesis procedures
3. English speaking

Exclusion Criteria:

1. Patients having microsurgical techniques as the primary procedure, such as an isolated laminotomy or microdiscectomy
2. Patients having surgery for spinal deformity as the primary indication
3. Patients having revision surgery
4. Patients having surgery for pseudarthrosis, trauma, infection, or tumor
5. Presence of back and/or lower extremity pain < 3 months
6. History of neurological disorder, resulting in moderate to severe movement dysfunction
7. Unable to provide stable address and access to internet and smartphone or tablet/iPad/computer/laptop indicating the inability to participate in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Mean daily post-operative physical activity as measured by an accelerometer. | Baseline to 12 months post-surgery
  Post-operative physical activity will be calculated as the average steps/day over a period of 7 days as measured by accelerometer

SECONDARY OUTCOMES:
Post-operative physical activity as measured by an accelerometer. | Baseline to 12 months post-surgery
  Post-operative physical activity will be calculated as the time spent in different intensities of physical activity over a period of 7 days as measured by accelerometer
Physical function as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) - Physical Function Domain | Baseline to 12 months post-surgery
  The PROMIS Physical Function 4-item short form will be used to measure physical function. Each item is measured from 1 to 5, representing low to high physical function, respectively. Total score ranges from 4 to 20. Total raw scores will be converted to T-scores.
Disability as measured by the Oswestry Disability Index. | Baseline to 12 months post-surgery
  The ODI has 10 items and scores range from 0 to 100%. A higher score represents higher disability.
Back pain as measured by the Numeric Rating Scale (NRS). | Baseline to 12 months post-surgery
  The NRS has 1 item and scores range from 0 to 10. A higher score represents more back pain.
Leg pain as measured by the Numeric Rating Scale (NRS). | Baseline to 12 months post-surgery
  The NRS has 1 item and scores range from 0 to 10. A higher score represents more leg pain.
Opioid Use as measured by patient self-report. | Baseline to 12 months post-surgery
  A single-item patient-reported opioid use question that ask about current opioid use.
Depression as measured by the Patient Reported Outcomes Measurement Information System (PROMIS) - Depression Domain | Baseline to 12 months post-surgery
  Depression 4-item short form will be used to measure depression. Responses for each item vary from Never, Rarely, Sometimes, Often, and Always. The lowest score is 4 and the highest score is 20, with higher scores indicating greater severity of depression.Total raw scores will be converted to T-scores.
Pain self-efficacy as measured by the Pain Self-Efficacy Questionnaire (PSEQ) | Baseline to 12 months post-surgery
  PSEQ has 10 items and responses vary from Not at all confident to completely confident. The lowest score is 0 and the highest score is 60 with a higher score representing higher pain self-efficacy.
Fear of movement as measured by theTampa Scale of Kinesiophobia. | Baseline to 12 months post-surgery
  The 17-item Tampa Scale of Kinesiophobia will be used to measure fear of movement. It has two sub-scales (activity avoidance and fear of pain) and the total score ranges from 17 to 68 with higher scores indicating greater fear of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Archer, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coronado RA, Master H, White DK, Pennings JS, Bird ML, Devin CJ, Buchowski MS, Mathis SL, McGirt MJ, Cheng JS, Aaronson OS, Wegener ST, Archer KR. Early postoperative physical activity and function: a descriptive case series study of 53 patients after lumbar spine surgery. BMC Musculoskelet Disord. 2020 Nov 27;21(1):783. doi: 10.1186/s12891-020-03816-y. PMID 33246446